CLINICAL TRIAL: NCT01734135
Title: Trial of Provider Notification for Patients With High B-type Natriuretic Peptide and no Imaging to Identify Unsuspected Heart Failure.
Brief Title: Provider Notification for High B-type Natriuretic Peptide Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Heidenreich, Investigator, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CHFQUERI-1101
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2016-04

CONDITIONS: Heart Failure
Keywords: B type natriuretic peptide; heart failure; cardiac imaging; quality of care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual care
- Clinical Reminder (Experimental): A note is sent to the primary care provider using the electronic medical record indicating the high BNP result and potential benefit of measurement of the left ventricular ejection fraction. A draft order is placed for an echocardiogram for the provider to accept or delete.
  Interventions: Other: Clinical Reminder

INTERVENTIONS:
Other: Clinical Reminder — A note is sent to the primary care provider using the electronic medical record indicating the high BNP result and potential benefit of measurement of the left ventricular ejection fraction. A draft order is placed for an echocardiogram for the provider to accept or delete.
  Arms: Clinical Reminder

SUMMARY:
This proposal examines use of a clinical reminder to the primary provider of patient with a high B type natriuretic peptide but no prior imaging.

Electrical Medical Record-based Intervention to Determine whether Clinical Reminders Improve Heart Failure Management in Patients with High BNP Values and Unknown LVEF.

DETAILED DESCRIPTION:
Rationale: B type natriuretic peptide is known to be elevated (> 100 pg/ml) in patients with heart failure. Furthermore, treatments are available to improve survival and reduce hospitalization if the left ventricular ejection fraction (LVEF) is < 40%. Accordingly, guidelines recommend an LVEF measure for patients with suspected heart failure. Prior work has demonstrated that patients with high BNP values do not always have a measure of left ventricular ejection.

Hypothesis: A reminder to patients with BNP and no imaging may prompt providers to order appropriate imaging potentially leading to 1) identification of unsuspected depressed ejection fraction and 2) more appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* BNP >= 200 pg/ml in last 2 months

Exclusion Criteria:

* Measure of LVEF in the last 12 months
* Last measure of LVEF < 40%

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Measurement of left ventricular ejection fraction | 6 months after randomization
  numerator: Measurement of left ventricular ejection fraction within 6 months of randomization.
  denominator: All randomized patients

SECONDARY OUTCOMES:
Identification of LVEF < 40% | 6 months following randomizaiton
  Numerator: number of patients identified with an LVEF< 40% Denominator: all randomized patients
Treatment of Low LVEF | 6 months following randomization
  Numerator: number of patients with an LVEF < 40% and treatment with either an angiotensin converting enzyme inhibitor, angiotensin receptor blocker or evidence based beta-blocker (carvedilol, metoprolol succinate, bisoprolol).
  Denominator: all randomized patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Heidenreich, MD, MS, Principal Investigator — VA Palo Alto HCS
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States